CLINICAL TRIAL: NCT06191887
Title: Phase 1a/1b Dose Escalation and Cohort Expansion Study of the Safety and Efficacy of B-Cell Activating Factor Receptor (BAFFR)-Based Chimeric Antigen Receptor T-Cells (MC10029) in Subjects With Relapsed or Refractory BAFFR-Expressing B-Cell Hematologic Malignancies
Brief Title: B-Cell Activating Factor Receptor (BAFFR)-Based Chimeric Antigen Receptor T-Cells With Fludarabine and Cyclophosphamide Lymphodepletion for the Treatment of Relapsed or Refractory B-cell Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC230807; NCI-2023-10077 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-004166 (Other: Mayo Clinic Institutional Review Board); MC230807 (Other: Mayo Clinic)
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: B-Cell Non-Hodgkin Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Recurrent Transformed Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Marginal Zone Lymphoma; Refractory Small Lymphocytic Lymphoma; Refractory Transformed Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Bendamustine Hydrochloride; Biopsy; Specimen Handling; Cyclophosphamide; fludarabine; Leukapheresis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (BARRF based chimeric antigen receptor T-cells) (Experimental): Patients undergo leukapheresis. Patients then receive cyclophosphamide IV, over 60 minutes and fludarabine IV over 30 minutes on day -5 to -3 or bendamustine IV over 10 minutes on days -4 and -3. Patients receive BAFFR based chimeric antigen receptor T-cells IV on day 0. Patients undergo echocardiography and MRI at screening, CT scan, PET scan, bone marrow biopsy/aspirate and blood sample collection throughout the study and tumor biopsy at progression.
  Interventions: Biological: Autologous BAFFR-targeting CAR T Cells; Drug: Bendamustine; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography; Drug: Fludarabine; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Autologous BAFFR-targeting CAR T Cells — Given IV
  Other Names: Autologous BAFFR-CAR T Cells; Autologous BAFFR-CAR-expressing T-cells
Drug: Bendamustine — Given IV
  Other Names: SDX-105
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow biopsy/aspirate
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase I trial tests safety, side effects and best dose of B-cell activating factor receptor (BAFFR)-based chimeric antigen receptor T-cells, with fludarabine and cyclophosphamide lymphodepletion, for the treatment of patients with B-cell hematologic malignancies that has come back after a period of improvement (relapsed) or that does not respond to treatment (refractory). BAFFR-based chimeric antigen receptor T-cells is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Giving chemotherapy, such as fludarabine and cyclophosphamide, helps ill cancer cells in the body and helps prepare the body to receive the BAFFR based chimeric antigen receptor T-cells. Giving BAFFR based chimeric antigen receptor T-cells with fludarabine and cyclophosphamide for lymphodepletion may work better for the treatment of patients with relapsed or refractory B-cell hematologic malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of (MC10029) autologous BAFFR-targeting chimeric antigen receptor (CAR) T cells following lymphodepleting (LD) therapy in subjects with relapsed or refractory BAFFR expressing B-cell hematologic malignancies.

II. To determine the recommended dose for phase 1b (dose expansion) and recommend phase 2 dose.

SECONDARY OBJECTIVES:

I. To assess the efficacy and antitumor activity of MC10029 in subjects with relapsed or refractory BAFFR-expressing B-cell hematologic malignancies.

II. To determine long-term toxicities in MC10029 recipients. III. To determine feasibility of manufacturing success rate of MC10029.

CORRELATIVE RESEARCH OBJECTIVES:

I. To evaluate the pharmacokinetics of MC10029 in peripheral blood samples. II. To study the relationship between BAFFR expression and clinical activity of MC10029.

OUTLINE:

Patients undergo leukapheresis. Patients then receive cyclophosphamide intravenously (IV), over 60 minutes and fludarabine IV over 30 minutes on day -5 to -3 or bendamustine IV over 10 minutes on days -4 and -3. Patients receive BAFFR based chimeric antigen receptor T-cells IV on day 0. Patients undergo echocardiography and magnetic resonance imaging (MRI) at screening, computed tomography (CT) scan, positron emission tomography (PET) scan, bone marrow biopsy/aspirate and blood sample collection throughout the study and tumor biopsy at progression.

After completion of study treatment, patients followed up at day 1, 2, 3, 4, 8, 11, 14, 21, 28, 60, 90, 180, 270, 365, 545 and 730 and then periodically for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION: Age ≥ 18 years
* PRE-REGISTRATION: Confirmed diagnosis of 1 of the following relapsed or refractory B-cell hematologic malignancies: chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), follicular lymphoma (FL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), or large B cell lymphoma (LBCL) including Richter's transformation from CLL/SLL

  * For CD19+ B cell malignancies; relapsed or refractory disease is defined by one of the following histopathology:

    * Biopsy proven SLL or flow cytometry proven CLL; relapsed or refractory disease is defined as:
    * Demonstration of progressive or stable disease by positron emission tomography/computed tomography (PET/CT) or computed tomography (CT) criteria according to the international workshop on chronic lymphocytic leukemia (iwCLL) 2018 criteria
    * Biopsy proven B-cell non-Hodgkin lymphoma (NHL) of any histopathology (including Richter Transformation of CLL); relapsed or refractory disease is defined as:
    * Demonstration of progressive or stable disease by PET/CT or CT criteria as the best response to the most recent chemotherapy regimen according to the revised Lugano Response Criteria for Malignant Lymphoma
* PRE-REGISTRATION: Disease Specific prior lines of therapies below:

  * For CLL/SLL, patients must have received ≥ two prior lines of therapy, and/or ≥ 6 months of second line prior BTK inhibition (e.g. ibrutinib or other such as acalabrutinib or zanubrutinib) and must have failed to respond to venetoclax or be intolerant. Exception: Patients in stable disease (SD) or partial response (PR) with a known ibrutinib resistance mutation (BTK or phospholipase Cγ2) may be included even if on ibrutinib therapy for less than 6 months

    * These patients may or may not have received prior antibody directed against cluster of differentiation 20 (CD20).
  * For Follicular Lymphoma, patients must have received ≥ two prior lines of therapy, including an antibody directed against CD20.

    * NOTE: Prior cluster of differentiation 19 (CD19) directed chimeric antigen receptor T-cell therapy (CART) must have a 100-day washout period.
  * For Mantle Cell Lymphoma, patients must have received ≥ two prior lines of therapy, including an antibody directed against CD20, and a BTK inhibitor.

    * NOTE: Prior CD19 directed CART must have a 100-day washout period.
  * For Marginal Zone Lymphoma, patients must have received ≥ two prior lines of therapy, including an antibody directed against CD20.

    * NOTE: Prior CD19 directed CART must have a 100-day washout period.
  * For Large B cell Lymphoma, patients must have received ≥ two prior lines of therapy, including an antibody directed against CD20. Prior exposure to CD19 directed CART will be allowed at the discretion of the Principal Investigator.

    * NOTE: Prior failed CD19 directed CART must have a 100-day washout period
  * For Richter's Transformation, patients must have received ≥two prior lines of therapy, including an antibody directed against CD20.
  * 100-day washout period starts from the date of the last prior CAR-T infusion.
* PRE-REGISTRATION: Measurable disease
* REGISTRATION: Positive BAFFR test
* REGISTRATION: Measurable disease
* REGISTRATION: Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* REGISTRATION: Hemoglobin ≥ 9.0 g/dL (unless due to documented marrow involvement with disease) obtained ≤14 days prior to registration
* REGISTRATION: Absolute neutrophil count (ANC) ≥ 1500/mm^3 (unless due to documented marrow involvement with disease) obtained ≤14 days prior to registration
* REGISTRATION: Platelet count ≥100,000/mm^3 (unless due to documented marrow involvement with disease) obtained ≤ 14 days prior to registration
* REGISTRATION: Total bilirubin ≤ 1.5 x upper limits of normal (ULN) (Subjects with Gilbert's Syndrome may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN) obtained ≤ 14 days prior to registration
* REGISTRATION: Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3 x ULN (≤ 5 x ULN for patients with liver involvement) obtained ≤ 14 days prior to registration
* REGISTRATION: Prothrombin time (PT)/international normalized ratio (INR) /activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy obtained ≤ 14 days prior to registration

  * Patients on a stable, maintenance regimen of anticoagulant therapy for ≥ 30 days prior to registration may have PT/INR measurements > 1.5 X ULN if, in the judgment of the investigator, the patient is suitable for the study
* REGISTRATION: Calculated creatinine clearance ≥45 ml/min using the Cockcroft-Gault formula obtained ≤ 14 days prior to registration
* REGISTRATION: Negative pregnancy test done ≤ 7 days prior to registration, for persons of childbearing potential only. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* REGISTRATION: Provide written informed consent understand and comply with protocol-required study procedures
* REGISTARTION: Patients must have an ejection fraction (EF) of ≥ 45%
* REGISTRATION: Patients must have pulse ox measurements of > 92% on room air
* REGISTRATION: Willingness to provide mandatory blood specimens for correlative research
* REGISTRATION: Willing to return to enrolling institution for study follow-up

Exclusion Criteria:

* PRE-REGISTRATION: Prior solid organ transplantation
* PRE-REGISTRATION: Unstable angina, clinically significant arrhythmia, or myocardial infarction ≤ 6 months of prior to pre-registration, or grade 3 or higher pericardial effusion at the time of pre-registration
* PRE-REGISTRATION: Prior anti-BAFF-R therapies
* PRE-REGISTRATION: Known contraindication to lymphodepleting (LD) chemotherapy
* PRE-REGISTRATION: Use of systemic antitumor therapy or investigational agent ≤ 14 days, prior to pre-registration
* PRE-REGISTRATION: Receiving any other investigational agent which would be considered as a treatment for the BAFF-R
* PRE-REGISTRATION: Autologous HCT ≤ 60 days prior to pre-registration
* PRE-REGISTRATION: Uncontrolled intercurrent non-cardiac illness including, but not limited to:

  * Previous or concurrent malignancy
  * Ongoing or active infection
  * Psychiatric illness/social situations
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy * Persons of childbearing potential who are pregnant or breastfeeding
  * Life Expectancy of < 6 weeks
  * Persons requiring systemic corticosteroids (>10 mg prednisone or equivalent per day) and/or other immunosuppressive therapy. Patients are allowed to use topical corticosteroids
  * Any other conditions that would limit compliance with study requirements
* PRE-REGISTRATION: Detectable malignant cells from cerebrospinal fluid (CSF) or magnetic resonance imaging (MRI) indicating brain metastases during screening, or a history of central nervous system (CNS) involvement by malignancy (CSF or imaging) with still active disease. Note: Patients with a history of CNS involvement resolving after treatment and without active disease will be considered eligible if other inclusion criteria are met
* PRE-REGISTRATION: History of a seizure disorder, major cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
* PRE-REGISTRATION: Radiation therapy ≤ 14 days prior to pre-registration
* PRE-REGISTRATION: Prior allogeneic hematopoietic stem cell transplant (HCT) in ≤ 6 months prior to pre-registration; patients with active graft versus host disease (GVHD) will not be eligible regardless of duration from prior allogeneic HCT
* PRE-REGISTRATION: Human immunodeficiency virus (HIV) positive patients
* PRE-REGISTRATION: Subjects with New York Health Association (NYHA) class III or greater heart failure
* REGISTRATION: Eligible for auto-HCT based on investigator judgement
* REGISTRATION: Presence of active bacterial, viral, or fungal infection that is uncontrolled, based on investigator judgment
* REGISTRATION: Patients with active hepatitis B or hepatitis C infections are excluded from the study. Patients who are documented to be HIV positive or proven HIV infection from testing are ineligible for the study. Infectious disease testing (HIV-1, HIV-2, hepatitis C virus (HCV) antibody and polymerase chain reaction (PCR), hepatitis B virus (HBV) surface antigen, HBV surface antibody, HBV core antibody) performed ≤ 45 days prior to registration may be considered for subject eligibility
* REGISTRATION: Previous or concurrent malignancy, except basal cell or squamous cell skin carcinoma, adequately resected and in situ carcinoma of cervix, or a previous malignancy that was completely resected and has been in remission for ≥ 5 years prior to registration
* REGISTRATION: Persons of childbearing potential who are pregnant or breastfeeding
* REGISTRATION: Life expectancy of < 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLT) | Up to 28 days after MC10029 (autologous B-cell activating factor receptor [BAFFR]-targeting chimeric antigen receptor [CAR] T cells product) infusion
  DLTs are defined per the protocol and assessed by the number of DLTs that occur during the DLT evaluation period and persist beyond the specified duration (relative to the time of onset, defined as within 28 days).
Incidence and severity of treatment emergent adverse events | Up to 15 years
  Defined as adverse events (AEs) that occur or worsen in severity on or after MC10029 product infusion.

SECONDARY OUTCOMES:
Overall response rate | Up to 15 years
  Will be estimated by the number of patients with an objective status of complete response (CR) or partial response (PR) by the positron emission tomography-computed tomography (PET-CT) based response criteria . Will be assessed according to Lugano criteria for lymphomas (follicular lymphoma [FL], mantle cell lymphoma [MCL], marginal zone lymphoma [MZL], large b-cell lymphoma [LBCL]) and International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 criteria for chronic lymphocytic leukemia (CLL).
Complete response rate | Up to 15 years
  Will be assessed according to Lugano criteria for lymphomas (FL, MCL, MZL, LBCL) and iwCLL 2018 criteria for CLL.
Duration of response | Up to 15 years
  Defined as the time from onset of response to progression or death due to any reason, whichever occurs earlier.
Progression free survival | Up to 15 years
  Defined as the time from initiation of treatment to the occurrence of disease progression or death.
Overall survival | Up to 15 years
  Defined as the time from treatment to death, regardless of disease recurrence.
Number of conforming versus nonconforming products | Up to 15 years
  Will be noted and reported. A conforming cell product product must have met all release criteria for infusion. No patient will receive a non-conforming product under this protocol, thus this endpoint will be evaluated by the Quality Assurance/Quality Control team.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Kharfan-Dabaja, M.D., M.B.A., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States